CLINICAL TRIAL: NCT00676091
Title: A Phase 3, Randomized, Active-Controlled, Double-Blind Trial Evaluating the Safety, Tolerability, and Immunogenicity of a 13-valent Pneumococcal Conjugate Vaccine in Healthy Infants Given With Routine Pediatric Vaccinations in Brazil
Brief Title: Study Evaluating 13-valent Pneumococcal Conjugate Vaccine in Healthy Infants in Brazil
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 6096A1-012
Record Dates: First submitted 2008-04-08; First posted 2008-05-12 (Estimated); Results first posted 2010-10-15 (Estimated); Last update posted 2011-08-08 (Estimated); Status verified 2011-08

CONDITIONS: Vaccines, Pneumococcal Conjugate Vaccine
Keywords: Pneumococcal conjugate vaccine
MeSH Terms: interventions — Heptavalent Pneumococcal Conjugate Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 13vPnC (Experimental): 13-valent pneumococcal conjugate vaccine (13vPnC) 0.5 milliliter (mL) dose administered intramuscularly (IM) at 2, 4, and 6 months of age (infant series) and 12 months of age (toddler dose).
  Interventions: Biological: 13-Valent Pneumococcal Conjugate Vaccine (13vPnC)
- 7vPnC (Active Comparator): 7-valent pneumococcal conjugate vaccine (7vPnC) 0.5 mL dose administered IM at 2, 4, and 6 months of age (infant series) and 12 months of age (toddler dose).
  Interventions: Biological: 7-Valent Pneumococcal Conjugate Vaccine (7vPnc)

INTERVENTIONS:
Biological: 13-Valent Pneumococcal Conjugate Vaccine (13vPnC)
  Arms: 13vPnC
Biological: 7-Valent Pneumococcal Conjugate Vaccine (7vPnc)
  Arms: 7vPnC

SUMMARY:
The purpose of this study will be to analyze 13-valent pneumococcal vaccine given to healthy infants in Brazil for safety and tolerability, and to determine the immune response to the vaccines.

ELIGIBILITY:
Inclusion criteria:

* Healthy 1 month old infants
* Available for the duration of the study and reachable by telephone
* Able to complete two blood drawing procedures during the study

Exclusion criteria:

* Previous vaccination, contraindication or history of allergic reaction to vaccine or vaccine components
* Bleeding disorder, immune deficiency or significant chronic or congenital disease
* Previous receipt of blood products or immune globulin

Ages: 28 Days to 54 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 354 (Actual)
Dates: Start 2008-04; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (3):
- Brazil (3):
  - Curitiba
  - Florianópolis
  - Sau Paulo

RESULTS

PARTICIPANT FLOW:
Period: Infant Series
Arm/Group | 13vPnC | 7vPnC
Started | 177 | 177
Vaccinated Dose 1 | 163 | 162
Vaccinated Dose 2 | 159 | 162
Vaccinated Dose 3 | 158 | 161
Completed | 157 | 159
Not Completed | 20 | 18
Not completed — Parent or legal guardian request | 10 | 8
Not completed — Protocol Violation | 6 | 3
Not completed — Adverse Event | 2 | 3
Not completed — Failed to return | 1 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Died prior to receiving 7vPnC | 0 | 1
Period: After Infant Series
Arm/Group | 13vPnC | 7vPnC
Started | 157 | 159
Completed | 156 | 156
Not Completed | 1 | 3
Not completed — Adverse Event | 0 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Failed to return | 1 | 1
Period: Toddler Dose
Arm/Group | 13vPnC | 7vPnC
Started | 156 | 156
Completed | 153 | 156
Not Completed | 3 | 0
Not completed — Failed to return | 2 | 0
Not completed — Parent or legal guardian request | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 13vPnC | 7vPnC | Total
Number analyzed (Participants) | 163 | 162 | 325
Age Continuous [Mean (Standard Deviation); unit: months] | 2.2 (0.2) | 2.2 (0.2) | 2.2 (0.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 76 | 165
  Male | 74 | 86 | 160

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Serotype Specific IgG Antibody Concentration ≥0.35 Micrograms Per Milliliter (Mcg/mL) in the 13vPnC Group Relative to 7vPnC Group 1 Month After the Infant Series
Description: Percentage of participants achieving predefined antibody threshold ≥0.35 mcg/mL along with the corresponding 95% confidence interval (CI) for the 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (serotypes 1, 3, 5, 6A, 7F, and 19A) are presented.
Time Frame: 1 Month after the infant series (7 Months of age)
Population: Evaluable immunogenicity population: treatments as randomized at all expected doses, blood drawn within specified timeframes, at least 1 valid and determinate assay result for proposed analysis, and no major protocol violations. N=number of participants with a determinate IgG antibody concentration to the given serotype.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 156 | 158
percentage of participants
  Common serotypes - serotype 4 | 100.0 [97.7 to 100.0] | 100.0 [97.7 to 100.0]
  Common serotypes - serotype 6B | 96.8 [92.7 to 99.0] | 95.6 [91.1 to 98.2]
  Common serotypes - serotype 9V | 98.7 [95.4 to 99.8] | 100.0 [97.7 to 100.0]
  Common serotypes - serotype 14 | 98.1 [94.5 to 99.6] | 97.5 [93.6 to 99.3]
  Common serotypes - serotype 18C | 97.4 [93.6 to 99.3] | 98.1 [94.5 to 99.6]
  Common serotypes - serotype 19F | 94.2 [89.3 to 97.3] | 98.7 [95.5 to 99.8]
  Common serotypes - serotype 23F | 96.8 [92.7 to 99.0] | 93.0 [87.8 to 96.5]
  Additional serotypes - serotype 1 | 99.4 [96.5 to 100.0] | 2.5 [0.7 to 6.4]
  Additional serotypes - serotype 3 | 87.1 [80.8 to 91.9] | 4.4 [1.8 to 8.9]
  Additional serotypes - serotype 5 | 98.7 [95.4 to 99.8] | 38.2 [30.4 to 46.4]
  Additional serotypes - serotype 6A | 97.4 [93.6 to 99.3] | 52.6 [44.4 to 60.6]
  Additional serotypes - serotype 7F | 100.0 [97.7 to 100.0] | 1.3 [0.2 to 4.6]
  Additional serotypes - serotype 19A | 99.4 [96.5 to 100.0] | 98.7 [95.4 to 99.8]

2. Primary Outcome: Percentage of Participants Achieving Antibody Level ≥5 Enzyme-linked Immunosorbent Assay (ELISA) Units Per mL (EU/mL) for Pertussis in the 13vPnC Group Relative to 7vPnC Group 1 Month After the Infant Series
Description: Percentage of participants achieving predefined antibody threshold ≥5 enzyme-linked immunosorbent assay (ELISA) units per mL (EU/mL) along with the corresponding 95% CI for concomitant antigen pertussis (pertussis toxoid [PT], filamentous hemagglutinin [FHA], and pertactin [PRN]) are presented.
Time Frame: 1 month after the infant series (7 months of age)
Population: Evaluable immunogenicity population. N=number of participants with a determinate antibody concentration to the given concomitant vaccine component.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 156 | 158
percentage of participants
  PT ≥5 EU/mL | 35.9 [28.4 to 44.0] | 32.3 [25.1 to 40.2]
  FHA ≥5 EU/mL | 70.1 [62.2 to 77.2] | 71.5 [63.8 to 78.4]
  PRN ≥5 EU/mL | 93.5 [88.5 to 96.9] | 96.2 [91.9 to 98.6]

3. Secondary Outcome: Percentage of Participants Achieving Serotype Specific IgG Antibody Concentration ≥0.35 Mcg/mL in the 13vPnC Group Relative to 7vPnC Group 1 Month After the Toddler Dose
Description: as for outcome 1
Time Frame: 1 month after the toddler dose (13 months of age)
Population: Evaluable immunogenicity population. N=number of participants with a determinate IgG antibody concentration to the given serotype.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 152 | 152
percentage of participants
  Common serotypes - serotype 4 | 100.0 [97.6 to 100.0] | 100.0 [97.6 to 100.0]
  Common serotypes - serotype 6B | 97.4 [93.4 to 99.3] | 98.7 [95.3 to 99.8]
  Common serotypes - serotype 9V | 100.0 [97.6 to 100.0] | 100.0 [97.6 to 100.0]
  Common serotypes - serotype 14 | 100.0 [97.6 to 100.0] | 99.3 [96.4 to 100.0]
  Common serotypes - serotype 18C | 99.3 [96.4 to 100.0] | 100.0 [97.6 to 100.0]
  Common serotypes - serotype 19F | 99.3 [96.4 to 100.0] | 98.7 [95.3 to 99.8]
  Common serotypes - serotype 23F | 98.7 [95.3 to 99.8] | 99.3 [96.4 to 100.0]
  Additional serotypes - serotype 1 | 100.0 [97.6 to 100.0] | 2.7 [0.7 to 6.7]
  Additional serotypes - serotype 3 | 92.1 [86.5 to 95.8] | 7.5 [3.8 to 13.0]
  Additional serotypes - serotype 5 | 100.0 [97.6 to 100.0] | 72.1 [63.9 to 79.4]
  Additional serotypes - serotype 6A | 100.0 [97.6 to 100.0] | 92.1 [86.5 to 95.8]
  Additional serotypes - serotype 7F | 100.0 [97.6 to 100.0] | 4.2 [1.5 to 8.8]
  Additional serotypes - serotype 19A | 100.0 [97.6 to 100.0] | 100.0 [97.6 to 100.0]

4. Secondary Outcome: Percentage of Participants Achieving Antibody Level ≥5 EU/mL for Pertussis in the 13vPnC Group Relative to 7vPnC Group 1 Month After the Toddler Dose
Description: Percentage of participants achieving predefined antibody threshold ≥5 EU/mL along with the corresponding 95% CI for concomitant antigen pertussis (pertussis toxoid [PT], filamentous hemagglutinin [FHA], and pertactin [PRN]) are presented.
Time Frame: 1 month after the toddler dose (13 months of age)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 152 | 152
percentage of participants
  PT ≥5 EU/mL | 50.7 [42.4 to 58.9] | 49.3 [41.1 to 57.6]
  FHA ≥5 EU/mL | 91.4 [85.8 to 95.4] | 88.8 [82.7 to 93.3]
  PRN ≥5 EU/mL | 99.3 [96.4 to 100.0] | 98.7 [95.3 to 99.8]

5. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-specified Local Reactions: Infant Series Dose 1 (2 Months of Age)
Description: Pre-specified local reactions were reported using an electronic diary. Tenderness was scaled as Any (tenderness present); Significant (present and interfered with limb movement). Swelling and redness were scaled as Any (swelling or redness present); Mild (0.5 centimeters [cm] to 2.0 cm); Moderate (2.5 to 7.0 cm); Severe (> 7.0 cm). Participants may be represented in more than 1 category.
Time Frame: Within 4 days after dose 1 (2 months of age)
Population: Safety population: all participants who received at least 1 dose of study vaccine. N=number of participants reporting yes for at least 1 day or no for all days.
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 145 | 156
percentage of participants
  Tenderness: Any | 60.0 | 59.4
  Tenderness: Significant | 14.0 | 12.8
  Swelling: Any | 13.9 | 15.0
  Swelling: Mild | 10.3 | 13.6
  Swelling: Moderate | 5.9 | 1.4
  Swelling: Severe | 0.0 | 0.0
  Redness: Any | 10.3 | 13.4
  Redness: Mild | 8.8 | 11.4
  Redness: Moderate | 2.9 | 2.1
  Redness: Severe | 0.0 | 0.0

6. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-specified Local Reactions: Infant Series Dose 2 (4 Months of Age)
Description: as for outcome 5
Time Frame: Within 4 days after dose 2 (4 months of age)
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 137 | 145
percentage of participants
  Tenderness: Any | 53.3 | 53.8
  Tenderness: Significant | 9.4 | 11.9
  Swelling: Any | 12.1 | 13.8
  Swelling: Mild | 10.5 | 10.0
  Swelling: Moderate | 2.4 | 3.9
  Swelling: Severe | 0.0 | 0.0
  Redness: Any | 9.3 | 12.4
  Redness: Mild | 9.3 | 11.6
  Redness: Moderate | 0.0 | 1.6
  Redness: Severe | 0.0 | 0.0

7. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-specified Local Reactions: Infant Series Dose 3 (6 Months of Age)
Description: as for outcome 5
Time Frame: Within 4 days after dose 3 (6 months of age)
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 134 | 134
percentage of participants
  Tenderness: Any | 48.1 | 47.4
  Tenderness: Significant | 10.9 | 8.8
  Swelling: Any | 14.6 | 9.7
  Swelling: Mild | 12.2 | 9.7
  Swelling: Moderate | 4.2 | 0.9
  Swelling: Severe | 0.0 | 0.0
  Redness: Any | 10.7 | 14.0
  Redness: Mild | 10.7 | 13.3
  Redness: Moderate | 0.8 | 0.9
  Redness: Severe | 0.0 | 0.0

8. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-specified Local Reactions: Toddler Dose (12 Months of Age)
Description: as for outcome 5
Time Frame: Within 4 days after toddler dose (12 months of age)
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 128 | 128
percentage of participants
  Tenderness: Any | 64.3 | 53.2
  Tenderness: Significant | 18.3 | 13.3
  Swelling: Any | 11.5 | 10.5
  Swelling: Mild | 8.1 | 8.7
  Swelling: Moderate | 5.3 | 3.9
  Swelling: Severe | 0.0 | 0.0
  Redness: Any | 13.3 | 8.7
  Redness: Mild | 12.4 | 7.8
  Redness: Moderate | 0.9 | 1.0
  Redness: Severe | 0.0 | 0.0

9. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-specified Systemic Events: Infant Series Dose 1 (2 Months of Age)
Description: Pre-specified systemic events (any fever ≥ 38 degrees Celsius [C], decreased appetite, irritability, increased sleep, and decreased sleep) were reported using an electronic diary. Participants may be represented in more than 1 category.
Time Frame: Within 4 days after dose 1 (2 months of age)
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 154 | 154
percentage of participants
  Fever ≥38 but ≤39 degrees C | 18.0 | 19.9
  Fever >39 but ≤40 degrees C | 0.0 | 0.7
  Fever >40 degrees C | 0.0 | 0.0
  Decreased appetite | 26.6 | 28.0
  Irritability | 80.3 | 77.9
  Increased sleep | 56.6 | 52.4
  Decreased sleep | 39.7 | 27.5

10. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-specified Systemic Events: Infant Series Dose 2 (4 Months of Age)
Description: as for outcome 9
Time Frame: Within 4 days after dose 2 (4 months of age)
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 145 | 157
percentage of participants
  Fever ≥38 but ≤39 degrees C | 23.8 | 23.0
  Fever >39 but ≤40 degrees C | 3.2 | 0.8
  Fever >40 degrees C | 0.0 | 0.0
  Decreased appetite | 33.8 | 29.6
  Irritability | 80.4 | 79.2
  Increased sleep | 32.8 | 38.7
  Decreased sleep | 25.8 | 36.0

11. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-specified Systemic Events: Infant Series Dose 3 (6 Months of Age)
Description: as for outcome 9
Time Frame: Within 4 days after dose 3 (6 months of age)
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 148 | 144
percentage of participants
  Fever ≥38 but ≤39 degrees C | 22.6 | 22.4
  Fever >39 but ≤40 degrees C | 4.2 | 3.5
  Fever >40 degrees C | 0.8 | 0.9
  Decreased appetite | 37.9 | 32.2
  Irritability | 76.9 | 71.2
  Increased sleep | 35.7 | 36.9
  Decreased sleep | 27.6 | 34.1

12. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-specified Systemic Events: Toddler Dose (12 Months of Age)
Description: as for outcome 9
Time Frame: Within 4 days after toddler dose (12 months of age)
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 136 | 133
percentage of participants
  Fever ≥38 but ≤39 degrees C | 31.0 | 29.9
  Fever >39 but ≤40 degrees C | 1.8 | 3.0
  Fever >40 degrees C | 0.9 | 0.0
  Decreased appetite | 33.3 | 39.0
  Irritability | 67.2 | 68.8
  Increased sleep | 30.8 | 24.1
  Decreased sleep | 22.7 | 20.6

ADVERSE EVENTS:
Time Frame: Baseline through 1 Month after last study vaccination (13 Months). Local reactions and systemic events assessed within 4 days of dose: Infant Series Dose 1=2 months of age; Dose 2=4 months of age; Dose 3=6 months of age; Toddler Dose=12 months of age.
Description: Safety population = all randomized subjects with at least 1 dose of study treatment. An Adverse Event (AE) term may be reported as both a serious and non-serious AE, but are distinct events. AE may = serious for 1 subject and = non-serious for another subject or subject may have experienced both a serious and non-serious episode of the same event.
Groups:
- Infant Series 13vPnC: 13-valent pneumococcal conjugate vaccine (13vPnC) 0.5 milliliter (mL) dose administered intramuscularly (IM) at 2, 4, and 6 months of age (infant series).
- Infant Series 7vPnC: 7-valent pneumococcal conjugate vaccine (7vPnC) 0.5 mL dose administered IM at 2, 4, and 6 months of age (infant series).
- After the Infant Series 13vPnC: 13-valent pneumococcal conjugate vaccine (13vPnC) 0.5 mL dose administered IM at 2, 4, and 6 months of age (infant series); assessment 1 month after the infant series (7 months of age).
- After the Infant Series 7vPnC: 7-valent pneumococcal conjugate vaccine (7vPnC) 0.5 mL dose administered IM at 2, 4, and 6 months of age (infant series); assessment 1 month after the infant series (7 months of age).
- Toddler Dose 13vPnC: 13-valent pneumococcal conjugate vaccine (13vPnC) 0.5 mL dose administered IM at 12 months of age (toddler dose).
  7-valent pneumococcal conjugate vaccine (7vPnC) 0.5 mL dose administered IM at 12 months of age (toddler dose).
  Other Adverse Events (non-serious events): the number affected (N) for non-systematic (non-solicited) Other Adverse Events N=69; systematic (solicited) Local Reactions N=81; systematic (solicited) Systemic Events N=84. Total N at Risk=155: 1 participant had no record of safety information during the Toddler dose period and was not included in the Safety population.
- Toddler Dose 7vPnC: 7-valent pneumococcal conjugate vaccine (7vPnC) 0.5 mL dose administered IM at 12 months of age (toddler dose).
  Other Adverse Events (non-serious events): the number affected (N) for non-systematic (non-solicited) Other Adverse Events N=64; systematic (solicited) Local Reactions N=67; systematic (solicited) Systemic Events N=86.
Arm/Group | Infant Series 13vPnC | Infant Series 7vPnC | After the Infant Series 13vPnC | After the Infant Series 7vPnC | Toddler Dose 13vPnC | Toddler Dose 7vPnC
Serious Adverse Events (participants affected / at risk) | 10/163 | 10/162 | 10/163 | 5/162 | 2/155 | 3/156
Other Adverse Events (participants affected / at risk) | 140/163 | 140/162 | 18/163 | 12/162 | 84/155 | 86/156
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Infant Series 13vPnC (N=163) | Infant Series 7vPnC (N=162) | After the Infant Series 13vPnC (N=163) | After the Infant Series 7vPnC (N=162) | Toddler Dose 13vPnC (N=155) | Toddler Dose 7vPnC (N=156)
Congenital hydrocephalus (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Intussusception (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 1 | 1 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 2 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0
Meningitis viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia primary atypical (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 2 | 2 | 0 | 2
Muscle abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Periorbital cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Tracheobronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Tracheobronchitis viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 1
Hypotonic-hyporesponsive episode (Nervous system disorders) | 1 | 3 | 0 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Grand mal convulsion (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Breath holding (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 1 | 1 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Infant Series 13vPnC (N=163) | Infant Series 7vPnC (N=162) | After the Infant Series 13vPnC (N=163) | After the Infant Series 7vPnC (N=162) | Toddler Dose 13vPnC (N=155) | Toddler Dose 7vPnC (N=156)
Anaemia (Blood and lymphatic system disorders) | 4 | 3 | 0 | 0 | 1 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Atrial septal defect (Congenital, familial and genetic disorders) | 1 | 1 | 0 | 1 | 0 | 0
Hydrocele (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0
Ventricular septal defect (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0
Congenital hydrocephalus (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 0
Glucose-6-phosphate dehydrogenase deficiency (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cerumen impaction (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 4 | 3 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 1 | 1 | 0 | 0 | 0 | 0
Strabismus (Eye disorders) | 0 | 2 | 0 | 0 | 0 | 0
Eye discharge (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 14 | 10 | 0 | 0 | 2 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 8 | 9 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 9 | 6 | 0 | 0 | 0 | 3
Abdominal pain (Gastrointestinal disorders) | 9 | 3 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 6 | 4 | 0 | 1 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 2 | 2 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 1
Abnormal faeces (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Intussusception (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Oral mucosal discolouration (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Regurgitation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 2 | 3
Pyrexia (General disorders) | 12 | 8 | 1 | 0 | 2 | 3
Injection site reaction (General disorders) | 4 | 2 | 0 | 0 | 0 | 0
Irritability (General disorders) | 2 | 4 | 0 | 0 | 0 | 0
Injection site pain (General disorders) | 1 | 2 | 0 | 0 | 0 | 0
Tenderness (General disorders) | 1 | 1 | 0 | 0 | 0 | 0
Hypothermia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Inflammation (General disorders) | 1 | 0 | 0 | 0 | 1 | 0
Injection site exfoliation (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Injection site induration (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Injection site scar (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Injection site swelling (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Oedema (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vaccination site erythema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vaccination site pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vaccination site reaction (General disorders) | 0 | 1 | 0 | 0 | 1 | 0
Allergy to anthropod sting (Immune system disorders) | 2 | 5 | 0 | 0 | 0 | 0
Milk allergy (Immune system disorders) | 1 | 1 | 1 | 0 | 0 | 0
Allergy to anthropod bite (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Food allergy (Immune system disorders) | 1 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 54 | 54 | 2 | 0 | 11 | 7
Nasopharyngitis (Infections and infestations) | 55 | 43 | 0 | 0 | 19 | 16
Gastroenteritis (Infections and infestations) | 11 | 12 | 1 | 0 | 1 | 1
Perineal infection (Infections and infestations) | 7 | 9 | 0 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 9 | 6 | 1 | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 2 | 12 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 5 | 5 | 0 | 1 | 1 | 0
Ear infection (Infections and infestations) | 5 | 2 | 0 | 0 | 3 | 1
Varicella (Infections and infestations) | 6 | 1 | 0 | 0 | 0 | 2
Exanthema subitum (Infections and infestations) | 3 | 3 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 3 | 3 | 0 | 0 | 2 | 2
Otitis media (Infections and infestations) | 3 | 3 | 0 | 0 | 2 | 3
Pneumonia (Infections and infestations) | 2 | 4 | 2 | 0 | 2 | 0
Tracheobronchitis (Infections and infestations) | 3 | 3 | 1 | 0 | 0 | 2
Viral rash (Infections and infestations) | 2 | 3 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 1 | 3 | 0 | 1 | 0 | 1
Bronchopneumonia (Infections and infestations) | 2 | 1 | 2 | 2 | 1 | 3
Conjunctivitis bacterial (Infections and infestations) | 1 | 2 | 0 | 0 | 0 | 1
Laryngitis (Infections and infestations) | 0 | 3 | 0 | 0 | 2 | 1
Pharyngitis (Infections and infestations) | 2 | 1 | 0 | 0 | 3 | 1
Sinusitis (Infections and infestations) | 3 | 0 | 0 | 0 | 0 | 1
Asymptomatic bacteriuria (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0
Conjunctivitis viral (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0
Impetigo (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0
Otitis media acute (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 6
Pneumonia primary atypical (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0
Pyoderma (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 2 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 2 | 0
Candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Conjunctivitis infective (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea infectious (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Herpangina (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Injection site abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Menigitis viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Pertussis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pharyngitis bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Roseola (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0
Skin bacterial infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 1 | 0 | 0 | 6 | 3
Viral diarrhoea (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Viral tonsillitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Muscle abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Periorbital cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Tracheobronchitis viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Hand-foot-and-mouth disease (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Tonsillitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 3 | 1 | 0 | 0 | 0 | 1
Traumatic brain injury (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0 | 0 | 0
Abnormal weight gain (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 1 | 1
Weight gain poor (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 1
Lactose intolerance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0 | 0 | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Hypotonic-hyporesponsive episode (Nervous system disorders) | 1 | 3 | 0 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Grand mal convulsion (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypokinesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Poor quality sleep (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Psychomotor skills impaired (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Breath holding (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 1
Pyelocaliectasis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 12 | 0 | 0 | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 5 | 5 | 2 | 1 | 2 | 6
Allergic cough (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 1 | 2 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2 | 0 | 0
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 7 | 4 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 3 | 0 | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 3 | 2 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 3 | 0 | 0 | 0 | 0
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 | 3 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 3 | 0 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0
Pityriasis alba (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Prurigo (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Heat rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hyperaemia (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pallor (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Tenderness (any) (Skin and subcutaneous tissue disorders) | 87/145 | 92/155 | 0/0 | 0/0 | 81/126 | 67/126 — Infant Series Dose 1 and Toddler Dose; tenderness (any)=present at site of vaccination
Tenderness (any) (Skin and subcutaneous tissue disorders) | 72/135 | 78/145 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; tenderness (any)=present at site of vaccination
Tenderness (any) (Skin and subcutaneous tissue disorders) | 63/131 | 63/133 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; tenderness (any)=present at site of vaccination
Tenderness (significant) (Skin and subcutaneous tissue disorders) | 19/136 | 18/141 | 0/0 | 0/0 | 21/115 | 14/105 — Infant Series Dose 1 and Toddler Dose; Tenderness (significant)=present and interfered with limb movement
Tenderness (significant) (Skin and subcutaneous tissue disorders) | 12/127 | 16/134 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Tenderness (significant)=present and interfered with limb movement
Tenderness (significant) (Skin and subcutaneous tissue disorders) | 13/119 | 10/114 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Tenderness (significant)=present and interfered with limb movement
Swelling (any) (Skin and subcutaneous tissue disorders) | 19/137 | 21/140 | 0/0 | 0/0 | 13/113 | 11/105 — Infant Series Dose 1 and Toddler Dose; Swelling (any)=present at site of vaccination
Swelling (any) (Skin and subcutaneous tissue disorders) | 15/124 | 18/130 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Swelling (any)=present at site of vaccination
Swelling (any) (Skin and subcutaneous tissue disorders) | 18/123 | 11/113 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Swelling (any)=present at site of vaccination
Swelling (mild) (Skin and subcutaneous tissue disorders) | 14/136 | 19/140 | 0/0 | 0/0 | 9/111 | 9/103 — Infant Series Dose 1 and Toddler Dose; Swelling (mild)=0.5 to 2.0 centimeters (cm)
Swelling (mild) (Skin and subcutaneous tissue disorders) | 13/124 | 13/130 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Swelling (mild)=0.5 to 2.0 cm
Swelling (mild) (Skin and subcutaneous tissue disorders) | 15/123 | 11/113 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Swelling (mild)=0.5 to 2.0 cm
Swelling (moderate) (Skin and subcutaneous tissue disorders) | 8/136 | 2/138 | 0/0 | 0/0 | 6/113 | 4/102 — Infant Series Dose 1 and Toddler Dose; Swelling (moderate)=2.5 to 7.0 cm
Swelling (moderate) (Skin and subcutaneous tissue disorders) | 3/124 | 5/128 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Swelling (moderate)=2.5 to 7.0 cm
Swelling (moderate) (Skin and subcutaneous tissue disorders) | 5/120 | 1/113 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Swelling (moderate)=2.5 to 7.0 cm
Swelling (severe) (Skin and subcutaneous tissue disorders) | 0/135 | 0/138 | 0/0 | 0/0 | 0/110 | 0/100 — Infant Series Dose 1 and Toddler Dose; Swelling (severe) >7.0 cm
Swelling (severe) (Skin and subcutaneous tissue disorders) | 0/123 | 0/128 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Swelling (severe) >7.0 cm
Swelling (severe) (Skin and subcutaneous tissue disorders) | 0/119 | 0/112 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Swelling (severe) >7.0 cm
Redness (any) (Skin and subcutaneous tissue disorders) | 14/136 | 19/142 | 0/0 | 0/0 | 15/113 | 9/103 — Infant Series Dose 1 and Toddler Dose; Redness (any)=present at site of vaccination.
Redness (any) (Skin and subcutaneous tissue disorders) | 12/129 | 16/129 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Redness (any)=present at site of vaccination
Redness (any) (Skin and subcutaneous tissue disorders) | 13/121 | 16/114 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Redness (any)=present at site of vaccination
Redness (mild) (Skin and subcutaneous tissue disorders) | 12/136 | 16/140 | 0/0 | 0/0 | 14/113 | 8/102 — Infant Series Dose 1 and Toddler Dose; Redness (mild)=0.5 to 2.0 cm
Redness (mild) (Skin and subcutaneous tissue disorders) | 12/129 | 15/129 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Redness (mild)=0.5 to 2.0 cm
Redness (mild) (Skin and subcutaneous tissue disorders) | 13/121 | 15/113 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Redness (mild)=0.5 to 2.0 cm
Redness (moderate) (Skin and subcutaneous tissue disorders) | 4/136 | 3/140 | 0/0 | 0/0 | 1/110 | 1/101 — Infant Series Dose 1 and Toddler Dose; Redness (moderate)=2.5 to 7.0 cm
Redness (moderate) (Skin and subcutaneous tissue disorders) | 0/123 | 2/128 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Redness (moderate)=2.5 to 7.0 cm
Redness (moderate) (Skin and subcutaneous tissue disorders) | 1/120 | 1/113 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Redness (moderate)=2.5 to 7.0 cm
Redness (severe) (Skin and subcutaneous tissue disorders) | 0/135 | 0/138 | 0/0 | 0/0 | 0/110 | 0/100 — Infant Series Dose 1 and Toddler Dose; Redness (severe) >7.0 cm
Redness (severe) (Skin and subcutaneous tissue disorders) | 0/123 | 0/128 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Redness (severe) >7.0 cm
Redness (severe) (Skin and subcutaneous tissue disorders) | 0/119 | 0/112 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Redness (severe) >7.0 cm
Fever ≥ 38 degrees Celsius [C] but ≤ 39 degrees C (General disorders) | 25/139 | 28/141 | 0/0 | 0/0 | 36/116 | 32/107 — Infant Series Dose 1 and Toddler Dose; Fever ≥ 38 degrees C but ≤ 39 degrees C
Fever ≥ 38 degrees C but ≤ 39 degrees C (General disorders) | 31/130 | 31/135 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Fever ≥ 38 degrees C but ≤ 39 degrees C
Fever ≥ 38 degrees C but ≤ 39 degrees C (General disorders) | 28/124 | 26/116 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Fever ≥ 38 degrees C but ≤ 39 degrees C
Fever > 39 degrees C but ≤ 40 degrees C (General disorders) | 0/135 | 1/138 | 0/0 | 0/0 | 2/110 | 3/100 — Infant Series Dose 1 and Toddler Dose; Fever > 39 degrees C but ≤ 40 degrees C
Fever > 39 degrees C but ≤ 40 degrees C (General disorders) | 4/124 | 1/128 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Fever > 39 degrees C but ≤ 40 degrees C
Fever > 39 degrees C but ≤ 40 degrees C (General disorders) | 5/119 | 4/113 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Fever > 39 degrees C but ≤ 40 degrees C
Fever > 40 degrees C (General disorders) | 0/135 | 0/138 | 0/0 | 0/0 | 1/110 | 0/100 — Infant Series Dose 1 and Toddler Dose; Fever > 40 degrees C
Fever > 40 degrees C (General disorders) | 0/123 | 0/128 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Fever > 40 degrees C
Fever > 40 degrees C (General disorders) | 1/119 | 1/112 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Fever > 40 degrees C
Decreased appetite (General disorders) | 38/143 | 40/143 | 0/0 | 0/0 | 39/117 | 46/118 — Infant Series Dose 1 and Toddler Dose; Decreased appetite
Decreased appetite (General disorders) | 44/130 | 40/135 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Decreased appetite
Decreased appetite (General disorders) | 50/132 | 39/121 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Decreased appetite
Irritability (General disorders) | 122/152 | 116/149 | 0/0 | 0/0 | 84/125 | 86/125 — Infant Series Dose 1 and Toddler Dose; Irritability
Irritability (General disorders) | 111/138 | 122/154 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Irritability
Irritability (General disorders) | 110/143 | 99/139 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Irritability
Increased sleep (General disorders) | 81/143 | 77/147 | 0/0 | 0/0 | 36/117 | 26/108 — Infant Series Dose 1 and Toddler Dose; Increased sleep
Increased sleep (General disorders) | 41/125 | 55/142 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Increased sleep
Increased sleep (General disorders) | 46/129 | 45/122 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Increased sleep
Decreased sleep (General disorders) | 56/141 | 38/138 | 0/0 | 0/0 | 27/119 | 22/107 — Infant Series Dose 1 and Toddler Dose; Decreased sleep
Decreased sleep (General disorders) | 33/128 | 49/136 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Decreased sleep
Decreased sleep (General disorders) | 35/127 | 43/126 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Decreased sleep

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.